CLINICAL TRIAL: NCT03037268
Title: Quality and Diagnostic Utility of Mydriatic Fundus Plenoptic Photography: The Plenoptic Ophthalmoscopy Reliability Trial
Brief Title: Quality and Diagnostic Utility of Mydriatic Fundus Plenoptic Photography
Acronym: PORT
Status: Withdrawn | Type: Observational
Why Stopped: Device is no longer available
Sponsor: Wills Eye (Other)
Collaborators: Mid Atlantic Retina (Other)
Responsible Party: Principal Investigator, Jason Hsu, MD, Dr., MD, Wills Eye
Other Study IDs: 14-447E
Record Dates: First submitted 2017-01-23; First posted 2017-01-31 (Estimated); Last update posted 2019-11-13 (Actual); Status verified 2019-11

CONDITIONS: Retinal Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients undergoing dilated examination: * examined in the Retina Service of Wills Eye Hospital
  * with and without visually significant posterior retinal or optic nerve pathology
  * imaged with a Lytro Plenoptic Camera and 28D lens
  Interventions: Device: Lytro Plenoptic Camera and 28D lens

INTERVENTIONS:
Device: Lytro Plenoptic Camera and 28D lens — * visual acuity measured, intraocular pressure obtained, eyes dilated as part of a standard exam for intended patient visit
  * screened and consented for study
  * subjected to bilateral plenoptic ophthalmoscopy
  * mydriatic, single-field fundus images obtained
  * images reviewed for quality and diagnostic utility by a masked grader

SUMMARY:
1. Establish the quality of fundus images produced by plenoptic ophthalmoscopy using the grading system proposed and utilized in the Fundus Photography versus Ophthalmoscopy Trials Outcomes in the Emergency Department (FOTO-ED) Study.
2. Determine diagnostic utility of plenoptic ophthalmoscopy images by comparing masked image reviewers' quality measurements and findings to images obtained with a commercially available ocular fundus camera and documented exam findings

DETAILED DESCRIPTION:
Visualization of the ocular fundus is considered an essential part of the physical examination, as abnormalities of the optic nerve, retinal vessels, and macula can reveal underlying systemic diseases and explain the etiology of visual complaints.

The Fundus Photography versus Ophthalmoscopy Trials Outcomes in the Emergency Department (FOTO-ED) Study demonstrated that only 14% of patients with complaints and conditions in which fundus examination is considered important had direct ophthalmoscopy performed by an ED physician .Greater than 80% of previously unknown fundus findings relevant to ED patient management were missed by ED physicians, but were identified by nonmydriatic digital fundus photography. Several of these cases resulted in recall of a discharged patient back to the ED for hospital admission once diagnostic fundus photos were reviewed.

In the search for an alternative to improve ease of use and fundus image quality, plenoptic technology provides a promising option for portable fundus imaging. Plenoptic, or light field, imaging has recently been introduced commercially with the release of the Lytro Plenoptic Camera (Mountain View, CA, USA). Utilizing an array of microlenses, the Lytro camera captures all available light in a scene from multiple vectors. By dividing up a scene as a whole with many individual microlenses, images can be refocused in post processing after acquisition, sharp focus can be attained in low light situations, and stereo images with perspective shifting can be attained.

To date there have been no published quantitative descriptions of the quality and reliability of plenoptic ophthalmoscopy using a commercially available, portable light field camera. Initial work from a pilot study using animal and human eyes was published in 2016. The purpose of the proposed prospective, cross sectional imaging study is to compare standard mydriatic fundus photography to a second generation camera developed with a Lytro plenoptic camera and customized light source, specifically analyzing diagnostic utility/sensitivity of detecting retinal pathology and overall image quality. If the image quality outcomes of the investigators proposed study are similar to those of the nonmydriatic fundus camera, the implications for physicians and the potential applications to ophthalmology related telemedicine are significant.

ELIGIBILITY:
Inclusion Criteria:

* With and without visually significant posterior retinal or optic nerve pathology,
* Pregnant women if already dilated for reason other than study participation.

Exclusion Criteria:

* Children,
* Prisoners,
* Poor view of posterior pole due to anterior segment pathology,
* Poor view of posterior pole due to posterior media opacities that necessitate use of B-scan ultrasound to evaluate posterior pole.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients undergoing dialted examination in the Retina Service of Wills Eye Hospital
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-12 (Estimated); Primary Completion 2019-05 (Estimated); Study Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
Image quality | through study completion, an average of 1 year
  Image quality grade (1 - 5, with 1 being excellent and 5 being not diagnostically useful)
Detection rate of "critical" retinal findings | through study completion, an average of 1 year
  Sensitivity (%) of detection of "critical" retinal findings with plenoptic ophthalmoscopy. Critical retinal findings include retinal detachment, retinal vascular sheathing, retinal hemorrhage, retinal whitening, optic disc edema, optic disc pallor, optic disc cupping (> 0.5 cup-to disc ratio)

CONTACTS AND LOCATIONS:
Overall Officials: Jason Hsu, MD, Principal Investigator — Wills Eye Hospital
Locations (1):
- Mid Atlantic Retina- Wills Eye Institute, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lamirel C, Bruce BB, Wright DW, Delaney KP, Newman NJ, Biousse V. Quality of nonmydriatic digital fundus photography obtained by nurse practitioners in the emergency department: the FOTO-ED study. Ophthalmology. 2012 Mar;119(3):617-24. doi: 10.1016/j.ophtha.2011.09.013. Epub 2012 Jan 3. PMID 22218140
- [Background] Bruce BB, Lamirel C, Wright DW, Ward A, Heilpern KL, Biousse V, Newman NJ. Nonmydriatic ocular fundus photography in the emergency department. N Engl J Med. 2011 Jan 27;364(4):387-9. doi: 10.1056/NEJMc1009733. No abstract available. PMID 21268749
- [Background] Adam MK, Aenchbacher W, Kurzweg T, Hsu J. Plenoptic Ophthalmoscopy: A Novel Imaging Technique. Ophthalmic Surg Lasers Imaging Retina. 2016 Nov 1;47(11):1038-1043. doi: 10.3928/23258160-20161031-08. PMID 27842198